CLINICAL TRIAL: NCT02317874
Title: A Phase 1 Study of Talazoparib (BMN 673) in Combination With Carboplatin and Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Testing the Addition of the Anti-Cancer Drug Talazoparib to the Combination of Carboplatin and Paclitaxel for the Treatment of Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02474; NCI-2014-02474 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 9782; 9782 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 9782 (Other: CTEP); UM1CA186716 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2014-12-17 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Carboplatin; Paclitaxel; Taxes; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schedule A (7-day talazoparib, paclitaxel, carboplatin) (Experimental): Patients receive talazoparib PO QD on days 1-7, paclitaxel IV over 1 hour on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  At any time after 4-6 cycles of treatment, patients may continue combination study therapy with talazoparib, carboplatin, and paclitaxel, talazoparib and carboplatin, talazoparib alone (continuous dosing), or observation without therapy at the discretion of the treating physician.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Talazoparib
- Schedule B (3-day talazoparib, paclitaxel, carboplatin) (Experimental): Patients receive talazoparib PO QD on days 1-3, paclitaxel IV over 1 hour on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  At any time after 4-6 cycles of treatment, patients may continue combination study therapy with talazoparib, carboplatin, and paclitaxel, talazoparib and carboplatin, talazoparib alone (continuous dosing), or observation without therapy at the discretion of the treating physician.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Talazoparib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase I trial studies the side effects and best dose of talazoparib when given together with carboplatin and paclitaxel in treating patients with solid tumors that have spread to other places in the body (advanced) or cannot be removed by surgery. Talazoparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving talazoparib with carboplatin and paclitaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of talazoparib (BMN 673) seven day schedule in combination with carboplatin and paclitaxel.

II. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of talazoparib (BMN 673) three day schedule in combination with carboplatin and paclitaxel.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity of talazoparib (BMN 673) in combination with carboplatin and paclitaxel.

II. To determine whether the pharmacokinetic parameters of talazoparib (BMN 673) when given in combination with carboplatin and paclitaxel correlate with thrombocytopenia.

III. To observe and record anti-tumor activity of talazoparib (BMN 673) alone after the combination with carboplatin, paclitaxel and talazoparib (BMN 673).

IV. To observe the safety and tolerability of talazoparib (BMN 673) in combination with paclitaxel and carboplatin and talazoparib (BMN 673) alone after the combination therapy.

EXPLORATORY OBJECTIVES:

I. To serially evaluate pharmacokinetic and pharmacodynamics parameters and use indirect pharmacokinetic/pharmacodynamics models to correlate with tumor response and resistance to the combination talazoparib (BMN 673), carboplatin, and paclitaxel therapy.

II. To explore mechanisms of resistance to the combination of talazoparib (BMN 673) with carboplatin and paclitaxel.

OUTLINE: This is a dose-escalation study of talazoparib. Patients are assigned to 1 of 2 dosing schedules.

SCHEDULE A: Patients receive talazoparib orally (PO) once daily (QD) on days 1-7, paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.

SCHEDULE B: Patients receive talazoparib PO QD on days 1-3, paclitaxel IV over 1 hour on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.

At any time after 4-6 cycles of treatment, patients may continue combination study therapy with talazoparib, carboplatin, and paclitaxel, talazoparib and carboplatin, talazoparib alone (continuous dosing), or observation without therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid malignancy (excluding lymphoma) that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective, and for which: a) there is reasonable expectation of response to the combination of carboplatin/paclitaxel OR b) BRCA 1/2 germline mutation is present; due to the longstanding acceptance of BRCA 1 and 2 mutation testing through Myriad, results from Myriad will be acceptable; if testing for BRCA 1 and 2 germline mutations is done through another organization, a report from a genetics consult with a qualified medical professional confirming that the laboratory results show a recognized germline deleterious BRCA 1 or 2 mutation or rearrangement is required; if the latter cannot be obtained, principal investigator (PI) or study chair review of the lab results and confirmation of BRCA mutation or rearrangement will be required OR c) BRCA 1/2 somatic mutation previously identified using a Clinical Laboratory Improvement Amendments (CLIA) certified assay
* Patients must have measurable or evaluable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 150,000/mcL
* Total bilirubin =< 1.25 x institutional upper limit of normal (ULN), with the exception of < 2.9 mg/dL for patients with Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN; =< 5 x ULN in setting of metastatic liver disease
* Creatinine =< 1.5 x upper limit of normal OR creatinine clearance >= 50 mL/min
* Ability to take oral medications
* Patients with central nervous system (CNS) metastases must be stable after therapy for CNS metastases (such as surgery, radiotherapy or stereotactic radiosurgery) for at least 4 weeks and must be off steroid treatment for 2 weeks prior to study enrollment
* The effects of talazoparib (BMN 673) on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of talazoparib (BMN 673) administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or targeted therapies within 2 weeks prior to entering the study or those who have not recovered (=< grade 1) from adverse events due to agents administered with the exception of any grade of alopecia
* No prior carboplatin unless given in neoadjuvant/adjuvant setting for curative intent and more than 6 months have elapsed since last carboplatin dose; in the case of relapsed ovarian cancer, patients are eligible if more than 6 months have elapsed since last carboplatin dose
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talazoparib (BMN 673) or other agents used in study
* Peripheral neuropathy of severity greater than grade 1
* The following medications are contraindicated or must be used with caution; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference

  * Contraindicated:

    * Cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) strong and moderate inhibitors
    * CYP2C8 inducers
    * Cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) strong and moderate inhibitors
    * CYP3A4 inducers
    * CYP3A4 sensitive substrates
  * Exclusions: the following supportive care medications will be allowed will be allowed as they are routinely administered with carboplatin and paclitaxel and have no potential interaction with talazoparib (BMN 673): dexamethasone, aprepitant, fosaprepitant, and ondansetron); oral pain medications such as hydrocodone, oxycodone taken on an as needed basis are also permitted
  * Transdermal products designed for systemic delivery must be assessed for interaction potential; topical products not designed to provide systemic delivery (including inhaled products, ophthalmologic products and transvaginal preparations) do not need to be considered since they do not have appreciable systemic absorption
  * Other contraindicated medications (per above) are not allowed unless close monitoring with labs or drug levels or by symptoms with subsequent dose adjustments is feasible; patients taking these concurrent medications are ineligible unless they can discontinue or switched to alternative medications prior to initiation of the study drug (at least 5 half-lives)
  * Use with caution:

    * CYP2C8 sensitive substrates
    * CYP2C8 weak inhibitors
    * CYP3A4 non-sensitive substrates
    * CYP3A4 weak inhibitors
  * These agents may be permitted if discontinuation is not feasible and no acceptable alternatives are available as determined by the treating physician; however, caution should be used; consider monitoring with labs or drug levels or by symptoms and consider dose adjustments of the medication
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because talazoparib (BMN 673) is a PARP inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with talazoparib (BMN 673), breastfeeding should be discontinued if the mother is treated with talazoparib (BMN 673); these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for interactions with study treatment; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* No clinically significant bleeding (i.e. gastrointestinal [GI] bleed, intracranial bleeding) within 6 months or major surgery within 4 weeks; minor surgeries (i.e. port placement, cataract surgery) are allowed within 2 weeks
* Anticoagulation and anti-platelet therapies are not permitted (this includes coumadin, low molecular weight heparins, factor Xa inhibitors, aspirin and non-steroidal anti-inflammatory drug [NSAIDS] or other medicines with similar effects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase 2 dose of talazoparib three day schedule | 21 days
  Defined as the highest safely tolerated dose where 0/6 or 1/6 (less than 33%) patients experience a dose-limiting toxicity and two or more patients have experienced a dose-limiting toxicity at the next higher dose level. Adverse events will be evaluated by type and severity using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 until March 31, 2018. CTCAE version 5.0 will be utilized beginning April 1, 2018. Adverse events data collection include adverse event diagnosis, date of onset and resolution, whether the event is ongoing, CTCAE grade, whether the event is serious, frequency, and outcome status, and action taken.
Maximum tolerated dose and recommended phase 2 dose of talazoparib seven day schedule | 21 days
  Defined as the highest safely tolerated dose where 0/6 or 1/6 (less than 33%) patients experience a dose-limiting toxicity and two or more patients have experienced a dose-limiting toxicity at the next higher dose level. Adverse events will be evaluated by type and severity using the National Cancer Institute CTCAE version 4.0 until March 31, 2018. CTCAE version 5.0 will be utilized beginning April 1, 2018. Adverse events data collection include adverse event diagnosis, date of onset and resolution, whether the event is ongoing, CTCAE grade, whether the event is serious, frequency, and outcome status, and action taken.

SECONDARY OUTCOMES:
Incidence of toxicity | Up to 4 weeks after last dose of treatment
  Graded according to NCI CTCAE version 4.0 until March 31, 2018. CTCAE version 5.0 will be utilized beginning April 1, 2018. Toxicities observed will be summarized in terms of types and severities for each schedule and dose level separately. The number and severity of toxicity incidents will be analyzed descriptively in tabular format. Comparisons between dose level arms will be performed using Fisher's exact test. Ninety percent confidence intervals for dose-limiting toxicity rates will be constructed for dose levels with 6 or more patients.
Anti-tumor response | Up to 4 weeks after last dose of treatment
  Will be determined by Response Evaluation Criteria in Solid Tumors criteria. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease, stratified by treatment schedule. 90% confidence intervals for the proportions of subjects with a confirmed anti-tumor response will be computed for dose levels with 6 or more patients. Exact logistic regression analysis will be performed to evaluate the dose-response relationship. Chi-square or Fisher's exact test will be used to compare responses between treatment schedules.
Pharmacokinetic parameters (area under the curve and concentration) in plasma samples | Pre-dose and 4 hours after talazoparib administration on days 1 and 3 or 7 (depending on assigned schedule) of cycle 1 and 0 and 4 hours on day 1 of all subsequent cycles
  All pharmacokinetic parameters will be summarized by treatment schedule dose level using standard descriptive statistics: means, medians, ranges, and standard deviations (if numbers and distribution permit). The Jonckheere-Terpstra trend test will be performed to determine the significance of the association between increasing dose level and each of the pharmacokinetic parameters within each treatment schedule. A Spearman rank correlation analysis will be performed to determine the relationship between actual dose administered and the pharmacokinetic parameters.

OTHER OUTCOMES:
Maximum concentration levels from plasma samples | Pre-dose, 2 hours, and 4 hours after talazoparib administration on days 1 and 3 or 7 (depending on assigned schedule) of cycle 1 and day 1 of cycle 1
  Maximum concentration levels will be summarized in terms of means, standard deviations and ranges. Linear mixed effects modeling with subject specific random effects will be performed to evaluate maximum concentration and plasma concentration collected on day 1 and day 3 predict changes in peripheral blood mononuclear cells. Furthermore, the empirical Bayesian approach will be utilized to incorporate pharmacokinetic data from other phase I studies of the agent to construct a pharmacokinetic population model.
Changes in peripheral blood mononuclear cell levels | Cycle 1 day 1 to cycle 2 day 1
  Changes in peripheral blood mononuclear cell levels from the cycle 1, day 1 (prior to first talazoparib dose) assessment to the cycle 1, day 3 or 7 and cycle 2, day 1 assessments will be evaluated using a two-sample t-test.
Changes in mutation status | Baseline to time of progression (up to 4 weeks after last dose of treatment)
  The number and frequency of mutation status changes from the baseline biopsy assessment to the biopsy obtained at the time of progression will be summarized in tabular format. The frequency of mutation status changes will be analyzed using a paired t-test or nonparametric Wilcoxon Signed Rank test. A negative binomial regression model will be utilized to account for the dose effect. The presence of individual mutations will be compared between the baseline and time of progression assessment using a paired McNemar's test. The Benjamini-Hochberg method will also be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Kari B Wisinski, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (3):
- United States (3):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- [Derived] Leal TA, Sharifi MN, Chan N, Wesolowski R, Turk AA, Bruce JY, O'Regan RM, Eickhoff J, Barroilhet LM, Malhotra J, Mehnert J, Girda E, Wiley E, Schmitz N, Andrews S, Liu G, Wisinski KB. A phase I study of talazoparib (BMN 673) combined with carboplatin and paclitaxel in patients with advanced solid tumors (NCI9782). Cancer Med. 2022 Nov;11(21):3969-3981. doi: 10.1002/cam4.4724. Epub 2022 Apr 8. PMID 35396812